CLINICAL TRIAL: NCT03039257
Title: Single, High Dose Vitamin A Replacement in Patients Undergoing Hematopoietic Stem Cell Transplantation and Its Role on MBI-LCBI Rates
Brief Title: Vitamin A Replacement in Patients Undergoing HSCT and Its Role on MBI-LCBI Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-5937
Record Dates: First submitted 2017-01-31; First posted 2017-02-01 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Hematopoietic Stem Cell Transplant
Keywords: hematopoietic stem cell transplant; vitamin a
MeSH Terms: interventions — Vitamin A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitamin A (Other): Participants receive single dose vitamin A supplementation prior to HSCT. A 3x3 dose escalation/de-escalation design will be used for this study.
  Interventions: Dietary Supplement: Vitamin A

INTERVENTIONS:
Dietary Supplement: Vitamin A — Dose administration will start with 2500 IU/kg with maximum dose of 250,000 IU orally.

SUMMARY:
The primary objective of this study is to establish that single dose vitamin A supplementation is feasible and safe in pediatric and young adult bone marrow transplant recipients until day +30 (± 7 days) after hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
The investigators' preliminary data suggest that low levels of vitamin A directly impact risk of mucosal barrier injury laboratory-confirmed bloodstream infection (MBI-LCBI), likely via decreased gut permeability, and they hypothesize supplemental vitamin A at the time of HSCT can reduce the risk of MBI-LCBI and gastrointestinal graft versus host disease (GI GVHD). A 3x3 dose escalation/de-escalation study design will be used to determine the safety and dosing required to maintain vitamin A levels in the upper quartile of normal range for age at day +30 (± 7 days) with single dose vitamin A supplementation prior to hematopoietic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing HSCT.

Exclusion Criteria:

* Vitamin A hypersensitivity or allergy.
* Age less than 1 year at time of transplant.
* Baseline pre-HSCT vitamin A levels higher than the upper quartile of normal range for age.
* Enteral feeding or medication intolerance.
* Pregnancy.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2018-01-17 (Actual); Study Completion 2018-03-28 (Actual)

PRIMARY OUTCOMES:
Vitamin A Level | 30 days after HSCT
  Vitamin A level will be measured 30 days after HSCT.

SECONDARY OUTCOMES:
Incidence of mucosal barrier injury laboratory-confirmed bloodstream infection (MBI-LCBI) | 100 days after HSCT
  Incidence of mucosal barrier injury laboratory-confirmed bloodstream infection (MBI-LCBI) 100 days after HSCT.

CONTACTS AND LOCATIONS:
Overall Officials: Stella Davies, MBBS, PhD, MRCP, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No